CLINICAL TRIAL: NCT03279250
Title: A Pre-Operative Study to Assess the Effects of Apalutamide Plus LHRH Agonist or Apalutamide Plus Abiraterone Acetate Plus LHRH Agonist for Six Months for Prostate Cancer Patients at High Risk for Recurrence
Brief Title: Apalutamide and Gonadotropin-Releasing Hormone Analog With or Without Abiraterone Acetate in Treating Participants With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0527; NCI-2018-01064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0527 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; Gonadotropin-Releasing Hormone; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (LHRHa, apalutamide) (Experimental): Participants receive gonadotropin-releasing hormone analog (leuprolide, goserelin, or triptorelin as determined by treating physician) IM once every 3 months and apalutamide PO QD. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning no less than 48 hours after completion of therapy, participants undergo radical prostatectomy.
  Interventions: Drug: Apalutamide; Biological: Gonadotropin-releasing Hormone Analog; Procedure: Radical Prostatectomy
- Arm B (LHRHa, apalutamide, abiraterone acetate) (Experimental): Participants receive gonadotropin-releasing hormone analog and apalutamide as in arm A, abiraterone acetate PO QD, and prednisone PO QD. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning no less than 48 hours after completion of therapy, participants undergo radical prostatectomy.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Biological: Gonadotropin-releasing Hormone Analog; Drug: Prednisone; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
  Arms: Arm B (LHRHa, apalutamide, abiraterone acetate)
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Biological: Gonadotropin-releasing Hormone Analog — Given IM
  Other Names: GnRH Agonist; GnRH Analog; Gonadotropin-Releasing Hormone Agonist; Gonadotropin-Releasing Hormone Analogue; LH-RH agonist; LH-RH Analogs; LHRH Agonist; luteinizing hormone-releasing hormone agonist; Luteinizing Hormone-Releasing Hormone Analog
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm B (LHRHa, apalutamide, abiraterone acetate)
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase II trial studies how well apalutamide and gonadotropin-releasing hormone analog with or without abiraterone acetate work in treating participants with prostate cancer prior to surgery. Apalutamide and abiraterone acetate may stop the growth of cancer cells either by killing the cells or by blocking some of the enzymes needed for cell growth. Hormone therapy, using gonadotropin-releasing hormone analog, may fight prostate cancer by lowering the amount of testosterone the body makes. Giving apalutamide, gonadotropin-releasing hormone analog, and abiraterone acetate may work better in treating participants with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of pathologic stage =< pT2N0 at prostatectomy for Group A (gonadotropin-releasing hormone analog [luteinizing hormone releasing hormone agonist (LHRHa)] plus apalutamide 240 mg orally [PO] daily for 6 months as preoperative therapy) and Group B (LHRHa plus apalutamide 240 mg PO daily plus abiraterone acetate 1000 mg PO daily and prednisone 5 mg PO once daily [QD] for 6 months as preoperative therapy).

SECONDARY OBJECTIVES:

I. To assess the tumor epithelium volume following treatment in groups A and B. II. To assess the rate of positive surgical margins in Group A and Group B. III. To assess the time to prostate specific antigen (PSA) recurrence (TTRPSA). IV. To assess the safety profile of the two treatment arms (apalutamide with and without abiraterone acetate and low dose prednisone) for six months in a preoperative setting.

EXPLORATORY OBJECTIVES:

I. Assessment of the steroid hormone metabolome in blood plasma and tissue by liquid chromatography tandem mass spectrometry.

II. Assessment of androgen signaling (canonical and non-canonical) and candidate pathways of resistance to androgen signaling inhibition by protein and ribonucleic acid (RNA) analysis.

III. Assessment of citrate intracellular tricarboxylic acid cycle (TCA) metabolite concentrations with liquid chromatography-tandem mass spectrometry (LCMS/MS).

IV. Proportion of patients who achieve pathological complete response (CR). V. Hyperpolarized 1-13C-pyruvate imaging at study entry and at 3 months in Arm A and Arm B.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants receive gonadotropin-releasing hormone analog (leuprolide, goserelin, or triptorelin as determined by treating physician) intramuscularly (IM) once every 3 months and apalutamide PO QD. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning no less than 48 hours after completion of therapy, participants undergo radical prostatectomy.

ARM B: Participants receive gonadotropin-releasing hormone analog and apalutamide as in arm A, abiraterone acetate PO QD, and prednisone PO QD. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning no less than 48 hours after completion of therapy, participants undergo radical prostatectomy.

After completion of study treatment, participants are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate with no histological variants (such as small cell, sarcomatoid, pure ductal cancer, transitional cell carcinoma).
* Patients may have received one prior depot injection of LHRH agonist or LHRH antagonist (degarelix) within 30 days prior to study entry. Patients who have received any other prior hormonal therapy or any chemotherapy for prostate cancer will be excluded. (Patients who have discontinued finasteride or dutasteride or testosterone supplement for at least 2 weeks will be allowed to enroll).
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol.
* Have signed an informed consent document indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study.
* Written authorization for use and release of health and research study information has been obtained.
* Pathology review at Monroe Dunaway (MD) Anderson (Note: if patient's prostate biopsy was not read at MD Anderson, it must be reviewed at the study site to confirm eligibility).
* Prostate biopsy. If previous biopsy has been performed within 3 months of screening, second biopsy procedure will not be required, if archival biopsies and at least one formalin fixed paraffin embedded biopsy tissue block containing tumor is available.
* The following tumor stage and Gleason scores: a) clinical >= stage T1c/T2 tumor with Gleason score >=8 b) clinical stage >= T2b tumor with Gleason score >= 7 and PSA > 10 ng/ml.
* Serum testosterone > 150 ng/dL. For patients treated up to 1 month of LHRH agonist, a testosterone measurement prior to the LHRH treatment will be used to determine eligibility, and must have been > 150 ng/dL. If no testosterone level is available from before LHRHa injection up to 30 days prior to study entry, the patient will be ineligible.
* Patient is suitable for prostatectomy.
* No evidence of metastatic disease as determined by imaging procedures.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Hemoglobin >= 9.0 g/dL independent of transfusion.
* Platelet count >= 100,000/uL.
* Absolute peripheral neutrophil count (ANC) > 1,000.
* Creatinine clearance >= 50 mL/min.
* Serum potassium >= 3.5 mmol/L.
* Serum bilirubin =< 1.5 x upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN.
* Serum albumin >= 3 g/dl.
* Able to swallow the study drug whole as a tablet.
* Patients must have normal coagulation profile and no history of substantial non-iatrogenic bleeding diathesis.
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken.
* Life expectancy of greater than 12 months.

Exclusion Criteria:

* Patients who have had any prior chemotherapy or radiotherapy for prostate cancer.
* Patients who have had > 1 LHRH agonist or antagonist depot injection or received depot injection > 30 days before study entry.
* Patients may not be receiving any other investigational agents.
* Patients may not be receiving the concomitant administration of any systemic therapy, biologic therapy, or other agents with anti-tumor activity against prostate cancer while the patients are on study.
* Patients with known metastatic prostate cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leuprolide acetate, abiraterone acetate, prednisone or apalutamide or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with apalutamide and abiraterone. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Avoid concomitant strong CYP3A4 inducers during abiraterone acetate treatment. If a strong CYP3A4 inducer must be co-administered, increase the abiraterone acetate dosing frequency.
* Avoid co-administration of abiraterone acetate with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, exercise caution and consider a dose reduction of the concomitant CYP2D6 substrate.
* Patients receiving medications known to lower the seizure threshold are ineligible unless discontinued or substituted at least 4 weeks prior to study entry. These include: 1) aminophylline/theophylline; 2) atypical antipsychotics (e.g., clozapine, olanzapine, risperidone, ziprasidone); 3) bupropion; 4) lithium; 5) pethidine; 6) phenothiazine antipsychotics (e.g., prochlorperazine (compazine), chlorpromazine, mesoridazine, thioridazine); 7) tricyclic and tetracyclic antidepressants (e.g., amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine).
* Chronically uncontrolled hypertension, defined conventionally as consistent systolic pressures above 170 or diastolic pressures above 110 despite anti-hypertensive therapy. Note that this is NOT a criterion related to particular blood pressure (BP) results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes. (for example doctor's visit related stress i.e. "white coat syndrome".
* Requirement for corticosteroids greater than the equivalent of 10 mg of prednisone daily for more than 2 weeks.
* Poorly controlled diabetes defined by hemoglobin A1C > 9.0 at screening.
* Active or symptomatic viral hepatitis or chronic liver disease.
* Known history of pituitary or adrenal dysfunction.
* Other malignancy, except non-melanoma skin cancer, that is active or has a >= 30% probability of recurrence within 12 months.
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
* Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens, ketoconazole, or estrogens (5-alpha reductase inhibitors allowed), or LHRH agonists/antagonists (Note: LHRH allowed if begun within 1 month of day 1).
* Prior systemic treatment with an azole drug within four weeks of cycle 1 day 1.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of cycle 1 day 1.
* Allergies, hypersensitivity, or intolerance to prednisone, LHRH analog or excipients of prednisone LHRH analog, abiraterone acetate and apalutamide.
* Previous use of abiraterone acetate or other investigational CYP17 inhibitor (e.g., TAK-700).
* Previous investigational antiandrogens (e.g., apalutamide, enzalutamide, BMS-641988).
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study.
* Patients unable to tolerate transrectal ultrasound.
* Anti-androgens (steroidal or non-steroidal) such as cyproterone acetate, flutamide, nilutamide, bicalutamide, etc. other than assigned study drug unless given for =< 4 weeks.
* Estrogens, progestational agents such as megestrol, medroxyprogesterone, diethylstilbestrol (DES), cyproterone, spironolactone > 50 mg/kg, etc. unless discontinued at least two weeks prior to randomization.
* Androgens such as testosterone, dehydroepiandrosterone (DHEA), etc. unless discontinued at least two weeks prior to randomization.
* Herbal products that may decrease PSA levels (e.g., saw palmetto) unless discontinued two weeks prior to randomization.
* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated.
* Severe hepatic impairment (Child-Pugh Class C).
* History of significant bleeding disorder unrelated to cancer, including: 1) diagnosed congenital bleeding disorders (e.g., von Willebrand's disease); 2) diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) of screening visit; 3) history of gastrointestinal (GI) bleeding within 3 months of screening visit requiring >= 2 units packed red blood cells.
* Clinically significant cardiovascular disease including: 1) myocardial infarction within 6 months of screening visit; 2) uncontrolled angina within 3 months of screening visit; 3) congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within three months of the Screening visit results in a left ventricular ejection fraction that is >= 50%. 4) history of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes). 5) prolonged corrected QT interval by the Fridericia correction formula (QTcF) on the screening electrocardiogram (ECG) > 470 msec. 6) history of Mobitz II second degree or third degree heart block without a permanent pacemaker in place. 7) hypotension (systolic blood pressure < 86 mmHg or bradycardia with a heart rate of < 50 beats per minute on the screening ECG, unless pharmaceutically induced and thus reversible (i.e. beta blockers).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Venkatesh N, Chauhan PK, Mukhida SS, Grewal K, Aparicio A, Pilie PG, Subudhi SK, Corn PG, Sachdeva A, Desai M, Siddiqui BA, Zurita AJ, Pain D, Gregg JR, Frigo DE, Logothetis CJ, Msaouel P, Koutroumpakis E, Hahn AW. Evaluating Clinical Tools to Monitor Cardiovascular Risk in Men With Prostate Cancer Receiving Hormone Therapy. JCO Oncol Pract. 2025 Nov 7:OP2500506. doi: 10.1200/OP-25-00506. Online ahead of print. PMID 41202201
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 86 participants signed consent, 18 participants were not randomized (10 screen failures, 3 Insurance complications, 5 consent withdrawn )
Period: Overall Study
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate) | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Full Range); unit: years] | 64 [54 to 75] | 62 [43 to 77] | 63 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 34 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Rate of Pathologic Stage =< pT2N0 at Prostatectomy
Description: The study will provide a point estimate and 95% confidence interval of the proportion of patients with pathologic stage =< pT2N0 at prostatectomy for each arm. Patient characteristics will be summarized using descriptive statistics for each arm.
Time Frame: At the time of radical prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
Number analyzed (Participants) | 32 | 31
Participants | 13 | 12

2. Secondary Outcome: Number of Participants With Incidence of Adverse Events
Description: Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Incidence of serious adverse events and 95% confidence interval will be provided overall as well as for each major affected organ category.
Time Frame: From screening up to 4 weeks post-surgery, an average of 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
Number analyzed (Participants) | 34 | 34
Participants
  Serious | 1 | 2
  Non Serious | 34 | 34

3. Secondary Outcome: Tumor Epithelium Volume in the Surgical Specimen
Description: Tumor volume will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Secondary categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: At the time of radical prostatectomy
Population: Tumor epithelium volume in the surgical specimen analysis is unavailable due to no data collected.
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Assessment of Positive Surgical Margins in the Surgical Specimen
Description: Presence of positive surgical margins will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Secondary categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: At the time of radical prostatectomy
Population: Assessment of positive surgical margins in the surgical specimen analysis is not available due to no data collected.
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Prostate Specific Antigen Recurrence (TTRPSA)
Description: TTRPSA will be summarized by Kaplan-Meier estimates and confidence intervals. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Secondary categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: From the date of randomization up to 4 weeks post-surgery
Population: Time to prostate specific antigen recurrence (TTRPSA) analysis is not available due to no data collected.
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Assessment of Steroid Hormone Metabolome in Blood Plasma and Tissue
Description: Steroid hormone metabolome in blood plasma and tissue will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Exploratory categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: At radical prostatectomy
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assessment of Protein and Ribonucleic Acid (RNA) Analysis Results
Description: Assessment of protein and RNA analysis results will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Exploratory categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: At radical prostatectomy
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Citrate Intracellular Tricarboxylic Acid (TCA) Cycle Metabolite Concentrations
Description: Citrate intracellular TCA cycle metabolite concentrations will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Exploratory categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: At radical prostatectomy
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Pathological Response
Description: Pathological response will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Exploratory categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: Up to 4 weeks post-surgery
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Hyperpolarized 1-13C-pyruvate Imaging Results
Description: Hyperpolarized 1-13C-pyruvate imaging results will be summarized descriptively and graphically. Comparisons between two the arms or patient subgroups will use a t-test or non-parametric alternative as indicated. Exploratory categorical endpoints will be summarized using proportions with 95% confidence intervals. Comparisons between the two arms will use a chi-square test or Fisher's exact if indicated.
Time Frame: Up to 4 weeks post-surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From screening up to 4 weeks post-surgery, an average of 7 months
Arm/Group | Arm A (LHRHa, Apalutamide) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate)
All-Cause Mortality (participants affected / at risk) | 1/34 | 1/34
Serious Adverse Events (participants affected / at risk) | 1/34 | 2/34
Other Adverse Events (participants affected / at risk) | 34/34 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (LHRHa, Apalutamide) (N=34) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate) (N=34)
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (LHRHa, Apalutamide) (N=34) | Arm B (LHRHa, Apalutamide, Abiraterone Acetate) (N=34)
ALT increase (Investigations) | 3 (5) | 8 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 21 (28) | 15 (19)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
AST increase (Investigations) | 4 (5) | 9 (14)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 11 (12) | 6 (7)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 9 (9) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (14) | 8 (8)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
HbA1c increased (Endocrine disorders) | 2 (2) | 2 (2)
TSH increased (Endocrine disorders) | 9 (11) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 30 (36) | 24 (27)
GERD (Gastrointestinal disorders) | 2 (2) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 2 (2)
Hot flashes (Vascular disorders) | 31 (40) | 25 (31)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (17) | 13 (15)
Hypertension (Vascular disorders) | 5 (6) | 9 (14)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 9 (11) | 2 (3)
Hypothyrodism (Endocrine disorders) | 3 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 10 (12) | 2 (2)
Irritability (General disorders) | 4 (5) | 2 (2)
Lipase increase (Investigations) | 7 (11) | 9 (17)
Lymphocyte count decrease (Investigations) | 2 (4) | 4 (4)
Memory impairment (Nervous system disorders) | 7 (7) | 4 (4)
ACTH increase (Metabolism and nutrition disorders) | 0 (0) | 6 (8)
Insulin increase (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
LDH increase (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Vitamin D decrease (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 3 (3)
Personality change (Psychiatric disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 7 (11)
Amylase increase (Investigations) | 4 (7) | 5 (13)
Weight loss (Investigations) | 2 (2) | 3 (5)
White blood cell decrease (Investigations) | 4 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03279250/Prot_SAP_000.pdf